CLINICAL TRIAL: NCT02786875
Title: The Effect of the Combination of Low Glycemic Index Diet, Exercise and Vitamin D on Breast Cancer Recurrence: DEDiCa Study
Brief Title: Diet, Exercise and Vitamin D in Breast Cancer Recurrence
Acronym: DEDiCa
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Cancer Institute, Naples (Other)
Collaborators: Unity Health Toronto (Other); University of Catania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DEDiCa; 2015-005147-14 (EudraCT Number)
Record Dates: First submitted 2016-05-06; First posted 2016-06-01 (Estimated); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Breast Cancer
Keywords: lifestyle; low glycemic index diet; exercise; vitamin D; breast cancer; Mediterranean diet
MeSH Terms: conditions — Breast Neoplasms; Motor Activity | interventions — Diet, Mediterranean

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (high intensity program): (Experimental): Diet: low glycemic index (GI) Mediterranean diet. All carbohydrate foods will be low GI choices (GI<70 on bread scale, e.g. legumes, pasta al dente, barley, oat, apples, oranges, berries, nuts) within a healthy Mediterranean diet (≥5 servings veg/fruit per day, ≤1 serving red meat+cold cuts/week, <7% SFA).
  Moderate physical activity: brisk walk of at least 30min per day (or approximately 5000 steps) more than the habitual physical activity.
  Vitamin D supplement (cholecalciferol) up to 4000 IU/day to reach blood levels of 60-80 ng/ml of 25(OH)D.
  Interventions: Other: low Glycemic Index Mediterranean diet; Behavioral: Moderate physical activity; Drug: high level Vitamin D
- Group B (lower intensity program) (Active Comparator): Diet: general recommendations for a healthy Mediterranean diet (≥5 servings veg/fruit per day, ≤1 serving red meat+cold cuts/week, <7% SFA).
  Basic physical activity: general recommendations to avoid sedentary behaviour. Vitamin D supplement (cholecalciferol) will be given only if vitamin D insufficiency is detected to reach blood levels of 30 ng/ml of 25(OH)D.
  Interventions: Other: Mediterranean diet; Behavioral: Basic physical activity; Drug: normal level Vitamin D

INTERVENTIONS:
Other: low Glycemic Index Mediterranean diet — All carbohydrate foods will be low GI choices (GI<70 on bread scale, e.g. legumes, pasta al dente, barley, oat, apples, oranges, berries, nuts) within a healthy Mediterranean diet (≥5 servings veg/fruit per day, ≤1 serving red meat+cold cuts/week, <7% SFA).
  Other Names: Arm A
  Arms: Group A (high intensity program):
Other: Mediterranean diet — General recommendations for a healthy Mediterranean diet (≥5 servings veg/fruit per day, ≤1 serving red meat+cold cuts/week, <7% SFA).
  Other Names: Arm B
  Arms: Group B (lower intensity program)
Behavioral: Moderate physical activity — Brisk walk of at least 30min per day (or approximately 5000 steps) more than the habitual physical activity.
  Arms: Group A (high intensity program):
Behavioral: Basic physical activity — General recommendations for physical activity
  Arms: Group B (lower intensity program)
Drug: high level Vitamin D — Vitamin D supplement (cholecalciferol) up to 4000 IU/day to reach normal blood levels of 60-80 ng/ml of 25(OH)D.
  Other Names: Dibase
  Arms: Group A (high intensity program):
Drug: normal level Vitamin D — Vitamin D (cholecalciferol) will be given only if vitamin D insufficiency is detected to bring blood levels up to normal ranges of 30ng/mL.
  Other Names: Dibase
  Arms: Group B (lower intensity program)

SUMMARY:
The purpose of this study is to reduce breast cancer recurrence and hence increase disease-free survival through a lifestyle program that includes a low glycemic diet, physical activity and vitamin D supplementation in women with breast cancer living in a Mediterranean country.

DETAILED DESCRIPTION:
The aim of this study is to reduce breast cancer recurrence and hence increase disease-free survival through either a high intensity or a lower intensity lifestyle program that includes low glycemic index diet, physical activity and supplementation with vitamin D, for 33 months, in women living in Italy who have been surgically treated for breast cancer (either late stage or early stage but highly proliferative) within the previous 12 months. The objectives of the study are: to determine if the high intensity program is more efficacious than the lower intensity program in: 1) reducing breast cancer recurrence and 2) improving glycemic, hormonal, cardiovascular and cancer-related epigenetic markers.

ELIGIBILITY:
Inclusion Criteria:

1. Women with primary diagnosis of histologically confirmed breast cancer (T1 with Ki67≥30%, T2, T3 without metastasis) within 12 months from diagnosis.
2. Age ≥ 30 and < 75 years.
3. Patients who are able to comprehend and are willing to sign the consent form and are able to adhere to the protocol including scheduled clinic visits and assigned treatment.

Exclusion Criteria:

1. Patients who do not possess the inclusion criteria for this study.
2. Patients with sarcoidosis or other granulomatous diseases or with hypercalcemia (Ca>11mg/dL).
3. Patients with any previous or current concomitant other malignant cancer.
4. Pregnant or lactating women.
5. Patients with AIDS diagnosis
6. Patients with severe renal insufficiency
7. Patients with kidney stones (nephrocalcinosis or nephrolithiasis)
8. Patients participating in other lifestyle clinical trials

Ages: 30 Years to 74 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 506 (Actual)
Dates: Start 2016-11-04 (Actual); Primary Completion 2020-10-10 (Actual); Study Completion 2023-12-15 (Estimated)

PRIMARY OUTCOMES:
Recurrence of disease at study end | 33 months
  Disease-free survival (DFS) calculated as the percentage of patients alive without

SECONDARY OUTCOMES:
Changes in glycemic markers | up to 33 months
  blood levels of glucose, glycated hemoglobin, insulin
Changes in hormonal markers | upt to 33 months
  insulin-like growth factor-1 (IGF-1), estradiol, testosterone, sex hormone binding globulin (SHBG)
Changes in cardiovascular risk factors | up to 33 months
  body weight, waist circumference, blood pressure, cholesterol, triglycerides, C-reactive protein
Changes in epigenetic factors | up to 33 months
  microRNA

CONTACTS AND LOCATIONS:
Overall Officials: Egidio Celentano, M.D., Principal Investigator — National Cancer Institute IRCCS Pascale Naples (Italy); Livia S Augustin, PhD, Principal Investigator — National Cancer Institute IRCCS Pascale Naples (Italy); Massimo Libra, M.D., Principal Investigator — University of Catania, Italy
Locations (7):
- Italy (7):
  - Centro Riferimento Oncologico, Aviano
  - Azienda Ospedaliera Cannizzaro, Catania
  - Clinica Mediterranea, Napoli
  - Istituto Nazionale Tumori Fondazione G. Pascale, Napoli
  - Ospedale dei Colli Monaldi, Napoli
  - Ospedale Evangelico Betania, Napoli
  - Ospedale San Vincenzo, Taormina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Augustin LS, Libra M, Crispo A, Grimaldi M, De Laurentiis M, Rinaldo M, D'Aiuto M, Catalano F, Banna G, Ferrau' F, Rossello R, Serraino D, Bidoli E, Massarut S, Thomas G, Gatti D, Cavalcanti E, Pinto M, Riccardi G, Vidgen E, Kendall CW, Jenkins DJ, Ciliberto G, Montella M. Low glycemic index diet, exercise and vitamin D to reduce breast cancer recurrence (DEDiCa): design of a clinical trial. BMC Cancer. 2017 Jan 23;17(1):69. doi: 10.1186/s12885-017-3064-4. PMID 28114909